CLINICAL TRIAL: NCT03628417
Title: Fázis II, randomizált, kettős Vak vizsgálat a bőr metasztázisok kezelésére kálcium elektroporációval
Brief Title: Confirmatory Trial in the Evaluation of Ca Electroporation for the Treatment of Cutaneous Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Szeged University (Other)
Responsible Party: Principal Investigator, Erika Kis, Principal Investigator, Assistant Professor, Szeged University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 032104/2016/OTIG
Record Dates: First submitted 2017-11-07; First posted 2018-08-14 (Actual); Results first posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Cutaneous Melanoma
Keywords: cutaneous metastases; calcium electroporation; bleomycin electroporation
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Intervention Model Description: This randomized double blinded phase II study is comparing the effect of calcium electroporation with ECT with bleomycin on patients with cutaneous metastases of any histology where the metastases are randomized by block randomization and are done separately in each patient.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- Calcium Electroporation (Experimental): Calcium
  Calcium chloride 220 mmol/L (9 mg/ml):
  * Tumor < 0.5 cm³ - 1 ml/cm³ tumor volume
  * Tumor > 0.5 cm³ - 0,5 ml/cm³ tumor volume Tumor volume = ab²π/6 (a = longest diameter, b = longest diameter perpendicular to "a")
  Interventions: Procedure: Calcium Electroporation
- Bleomycin based electrochemotherapy (Experimental): Bleomycin
  Bleomycin 1000 IU/ml:
  * Tumor < 0.5 cm³ - 1 ml/cm³ tumor volume
  * Tumor > 0.5 cm³ - 0,5 ml/cm³ tumor volume Tumor volume = ab²π/6 (a = longest diameter, b = longest diameter perpendicular to "a")
  Maximum of injected bleomycin per tumor will be 1500 IU and total dose per treatment 7500 IU. Normal maximum limit for bleomycin is 15.000 IU/m² body surface area.
  Interventions: Procedure: Bleomycin based electrochemotherapy

INTERVENTIONS:
Procedure: Calcium Electroporation — If the patient agrees biopsies will be performed from the tumor area before and after electroporation during local anaesthesia. Maximum of 8 biopsies will be done, depending on the patient's number of metastases.
  All patient's regardless of the number of metastases will have one biopsy from area treated with calcium and one from area treated with bleomycin, after the randomization code is revealed at day 180.
  Patients with more than 6 metastases: One to two biopsies before treatment, one to two biopsies one week after treatment from metastases treated with calcium and bleomycin respectively.
  All biopsies will be handled according to current guidelines and analyzed by a pathologist for amount of tumor tissue, inflammation, fibrosis and necrosis.
  Arms: Calcium Electroporation
Procedure: Bleomycin based electrochemotherapy — If the patient agrees biopsies will be performed from the tumor area before and after electroporation during local anaesthesia. Maximum of 8 biopsies will be done, depending on the patient's number of metastases.
  All patient's regardless of the number of metastases will have one biopsy from area treated with calcium and one from area treated with bleomycin, after the randomization code is revealed at day 180.
  Patients with more than 6 metastases: One to two biopsies before treatment, one to two biopsies one week after treatment from metastases treated with calcium and bleomycin respectively.
  All biopsies will be handled according to current guidelines and analyzed by a pathologist for amount of tumor tissue, inflammation, fibrosis and necrosis.
  Arms: Bleomycin based electrochemotherapy

SUMMARY:
Electroporation is a method that can facilitate transport of molecules across the cell membrane and into the cell by means of electrical pulses. The method can be used with molecules that normally have difficulty passing the cell membrane such as chemotherapy (electrochemotherapy). Electrochemotherapy (ECT) is used in cancer therapy, where chemotherapy is administered intratumoral or intravenous, then followed by electrical pulses applied directly on the tumor. The chemotherapy accumulates in the cancer cells which results in an increased cytotoxic effect. The most used chemotherapeutic drug used in electrochemotherapy is bleomycin. Electrochemotherapy is a well-documented local treatment form for especially cutaneous tumors. Today, the treatment is used mostly in palliative care in more than 140 centres around Europe.

In vitro and in vivo studies have shown that the combination of calcium and electroporation is an effective method in killing cancer cells without serious side effects.This new combination opens the possibility of replacing bleomycin with calcium in treatments with electroporation.

Calcium electroporation is a local treatment where calcium is administered intratumoral and followed by electrical pulses applied on the tumor.

The preclinical studies have shown that there is a difference in sensitivity in tumor cells and normal cells, as normal cells tolerate the treatment better than tumor cells (own data manuscript in preparation). The studies have also shown that there is no cell injury by calcium injection without electroporation, the investigators therefore expect that the treatment only will cause minor side effects.

Calcium electroporation would be possible to use on patients for whom chemotherapy is contradicted e.g. severe lung functions impairment, pregnant woman etc. Calcium electroporation is a simple and unexpensive cancer treatment that does not involve any administration of cytotoxic chemotherapy, and can be performed by surgeons, radiologists as well as oncologists. Both electroporation equipment and calcium are already being used in the clinic, so the treatment can easily be implemented.

DETAILED DESCRIPTION:
Trial Design for Treatment of Cutaneous Metastases:

The current study is a randomized double blinded phase II study comparing the effect of calcium electroporation with ECT with bleomycin on patients with cutaneous metastases of any histology. As calcium and bleomycin are administered intratumoral, only small metastases from 0.5-3 cm will be treated. The treatments will be compared in tumor response and adverse events. Treatment will be done in a palliative purpose.

Cancer patients with cutaneous involvement have often several metastases. A maximum of ten metastases will be included per patient. One to six metastases (depending on the patient's number of metastases) will be numbered 1-6 and randomized into one of two treatment arms

1. Intratumoral calcium followed by electroporation
2. Intratumoral bleomycin followed by electroporation Randomization will be performed separately on each metastasis, so the patient may receive both treatments. Calcium and bleomycin will be mixed into syringes labeled with numbers according to the metastases and both treating doctor and patient will be blinded to the content of the syringes.

If the patient has more than six metastases, then one to four metastases will be used for biopsy. The treatment of these metastases will be known, and biopsies will be performed before and after treatment.

Biopsies will only be performed if the patient has more than six metastases. The metastases used for biopsy will not be evaluated on response.

The treatment will be performed in local or general anesthesia depending on location and number of metastases. Bleomycin/calcium will be administered intratumorally and immediately after the electrode will be placed on the metastasis. The electric pulses are generated using a cliniporator according to ESOPE (European Standard Operating Procedure of Electrochemotherapy). The therapy is a once only treatment and the patients will be followed up with regular clinical controls for six months. At follow up six months after treatment, the randomization code for the one patient will be revealed. If the patient agrees, biopsies will then be taken from an area treated with calcium and an area treated with bleomycin. Last visit will be one year after treatment.

To identify the metastases at follow up visits, the metastases will be marked with a pen, numbered and documented with clinical photos at baseline.

Randomization The metastases are randomized by block randomization and are done separately in each patient. The randomization is performed by an extern unit, using the computer program nQuery Adviser 7.0. The bleomycin and calcium are mixed and labeled by an extern unit, and since both calcium and bleomycin are transparent and identical in volume, it is possible to label the syringes in a manner to blind the treating doctor. The syringes are labeled with numbers according to the metastases so syringe number "1" goes to metastasis number "1" and so on. The randomization code is kept behind locked doors, and is not accessible to the treating doctor. The randomization code is revealed for each patient after follow up, 6 months after treatment.

The randomization code can be revealed before completion of the investigation, if the investigator believes that the treatment causes so serious unexpected events or reactions, that a continuation of treatment is unacceptable.

As the randomization is done separately in each patient, code-break is possible for the individual patient, without breaking the code of the other participants.

Dose In the preclinical study, the tumors were treated with isotonic calcium chloride solution 168 mmol/L and with a volume equivalent to 0.5 x tumor volume, and this with good effect. In another preclinical study the investigators have tested the effect of this dose in different tumor types and saw variable results of the response rate. Some tumor types showed slightly lower response at this dose (own data, manuscript in preparation). Because of this experience the investigators have decided to increase the dose of calcium chloride, in this trial, to 220 mmol/L.

Volume of calcium chloride is dependent on tumor volume. Smaller tumors should have bigger volume per cm³, as smaller tumors are expected to have a bigger loss of injected medicine into the surrounding tissue. The dose volume is calculated according to the "European Standard Operating Procedure of the Electrochemotherapy (ESOPE)".

Calcium

Calcium chloride 220 mmol/L (9 mg/ml):

* Tumor < 0.5 cm³ - 1 ml/cm³ tumor volume
* Tumor > 0.5 cm³ - 0.5 ml/cm³ tumor volume Tumor volume = ab2π/6 (a = longest diameter, b = longest diameter perpendicular to "a")

Bleomycin Both dose and volume of bleomycin is standard according to ESOPE

Bleomycin 1000 IU/ml:

* Tumor < 0.5 cm³ - 1 ml/cm³ tumor volume
* Tumor > 0.5 cm³ - 0,5 ml/cm³ tumor volume Tumor volume = ab²π/6 (a = longest diameter, b= longest diameter perpendicular to "a")

Maximum of injected bleomycin per tumor will be 1500 IU and total dose per treatment 7500 IU. Normal maximum limit for bleomycin is 15.000 IU/m² body surface area.

Bleomycin and calcium chloride are mixed and labeled according to current guidelines. The mixtures will be used in a maximum of 6 hours after mixing.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Verified cutaneous metastases of any histology.
* At least one cutaneous metastases between 0.5 to 3 cm and accessible to electroporation.
* The patient should have been offered current standard treatment. If there is no further standard treatment to offer, or if the patient does not want to receive this, the patient may be included in the trial.
* Treatment free interval of more than two weeks. However, patients treated with Navelbine (Vinorelbine) Capecitabine (Xeloda) or weekly paclitaxel (Taxol) can continue these treatments, if there is no regression of cutaneous metastases. Other medical cancer treatments such as endocrine treatment, targeted treatment and radiotherapy to another area may also continue.
* Performance status World Health Organization (WHO) ≤ 2.
* Expected survival of > 3 months.
* Platelets ≥ 50 billion/L, international normalized ratio (INR) < 1.5. Medical correction is allowed, e.g. correction of a high INR using vitamin K.
* Sexually active men and women who can become pregnant should use adequate contraception during this trial (pill, spiral, injection of prolonged progestin, subdermal implantation, hormone-containing vaginal devices, transdermal patches).
* The patient should be able to understand the information.
* Signed informed consent.

Exclusion Criteria:

* Previous bleomycin treatment with more than 200,000 U/m² .
* History of severe allergic reactions associated with bleomycin.
* Coagulation disorder which cannot be corrected.
* Pregnancy and lactation.
* Participating in other clinical trials involving experimental drugs or involved in a trial within 4 weeks prior to study drug administration.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2019-06-04 (Actual); Study Completion 2019-06-04 (Actual)

REFERENCES:
- [Background] Falk H, Forde PF, Bay ML, Mangalanathan UM, Hojman P, Soden DM, Gehl J. Calcium electroporation induces tumor eradication, long-lasting immunity and cytokine responses in the CT26 colon cancer mouse model. Oncoimmunology. 2017 Mar 17;6(5):e1301332. doi: 10.1080/2162402X.2017.1301332. eCollection 2017. PMID 28638724
- [Derived] Agoston D, Baltas E, Ocsai H, Ratkai S, Lazar PG, Korom I, Varga E, Nemeth IB, Dosa-Racz Viharosne E, Gehl J, Olah J, Kemeny L, Kis EG. Evaluation of Calcium Electroporation for the Treatment of Cutaneous Metastases: A Double Blinded Randomised Controlled Phase II Trial. Cancers (Basel). 2020 Jan 10;12(1):179. doi: 10.3390/cancers12010179. PMID 31936897
- See also: Calcium electroporation for treatment of cutaneous metastases; a randomized double-blinded phase II study, comparing the effect of calcium electroporation with electrochemotherapy — http://dx.doi.org/10.1080/0284186X.2017.1355109

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with cutan metastases of melanoma malignum and breast cancer were followed-up at one of the academic medical center in Hungary between September 2016 and June 2019 based on oncologist refferal.
Pre-assignment Details: Enrolled participants were not excluded from the study before assignment to groups. Block randomization was performed separately on each metastasis, so the patients received both treatments.
  The bleomycin and calcium syringes were mixed and labeled with numbers according to the metastases.
Units Other Than Participants: cutan metastases
Groups:
- Calcium Electroporation: Volume of calcium chloride (220 mmol/L) was dependent on tumor volume. Smaller tumors should have bigger volume per cm³, as smaller tumors were expected to have a bigger loss of injected medicine into the surrounding tissue.The dose volume was calculated according to the 'European Standard Operating Procedure of the Electrochemotherapy'.
  * Tumor < 0.5 cm³ - 1 ml/cm³ tumor volume
  * Tumor > 0.5 cm³ - 0,5 ml/cm³ tumor volume Tumor volume = ab²π/6 (a = longest diameter, b = longest diameter perpendicular to "a") Biopsies were performed from the tumor area before and after electroporation. Maximum of 8 biopsies were done, depending on the patient's number of metastases. All patient's regardless of the number of metastases had one biopsy from area treated with calcium and one from area treated with bleomycin, after the randomization code was revealed at day 180.
  All biopsies were handled and analyzed by a pathologist for amount of tumor tissue, inflammation, fibrosis and necrosis.
- Bleomycin Based Electrochemotherapy: Both dose and volume of bleomycin (1000 IU/ml) was standard according to ESOPE.
  * Tumor < 0.5 cm³ - 1 ml/cm³ tumor volume
  * Tumor > 0.5 cm³ - 0,5 ml/cm³ tumor volume Tumor volume = ab²π/6 (a = longest diameter, b = longest diameter perpendicular to "a") Maximum of injected bleomycin per tumor was 1500 IU and total dose per treatment was 7500 IU.
  Biopsies were performed from the tumor area before and after electroporation. Maximum of 8 biopsies were done, depending on the patient's number of metastases. All patient's regardless of the number of metastases had one biopsy from area treated with bleomycin and one from area treated with calcium, after the randomization code was revealed at day 180.
  All biopsies will be handled according to current guidelines and analyzed by a pathologist.
Period: Overall Study
Arm/Group | Calcium Electroporation | Bleomycin Based Electrochemotherapy
Started (If the patient has more than six metastases, then one to four metastases were used for biopsy.) | 7; 24 cutan metastases | 7; 20 cutan metastases
Day 0 (The treatment of the previously removed metastases (before and after treatment) were known.) | 7; 21 cutan metastases | 7; 17 cutan metastases
Day 7 | 7; 18 cutan metastases | 7; 15 cutan metastases
Day 15 | 7; 18 cutan metastases | 7; 15 cutan metastases
Day 30 | 7; 18 cutan metastases | 7; 15 cutan metastases
Day 60 | 7; 18 cutan metastases | 7; 15 cutan metastases
Day 90 | 7; 18 cutan metastases | 7; 15 cutan metastases
Day 180 (The randomization code was revealed for each patient. Biopsies were taken from both arms.) | 7; 12 cutan metastases | 7; 9 cutan metastases
Completed (The patients were followed a year after treatment.) | 6; 7 cutan metastases (One patient died and 3 more Ca electroporated lesions were removed before the one-year closing visit) | 6; 7 cutan metastases (One patient died before the one-year closing visit,this is why decreased the number of metastases)
Not Completed | 1; 17 cutan metastases | 1; 13 cutan metastases
Not completed — Death | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All participants receiving Calcium Electroporation and Bleomycin Based Electrochemotherapy.
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
Age, Customized [Median (Full Range); unit: years]
  Age | 70 [49 to 83]
Sex/Gender, Customized [Number; unit: Participants]
  Female | 5
  Male | 2
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 7
Patients with cutaneous metastases [Number; unit: Participants]
  Patients with MM cutaneous metastases | 6
  Patients with breast cc. cutaneous metastases | 1

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (RECIST1.1) of Calcium Electroporation and Bleomycin Based Electrochemotherapy on Cutaneous Metastases at Day 180.
Description: Documentation was done with digital color photography, including a ruler to estimate tumor size. Primary evaluation of the response was based on criteria similar RECIST 1.1 guidelines and defined as complete response (CR) - disappearance of the lesion, partial response (PR) - at least 30% decrease in the largest diameter of the lesion, progressive disease - at least 20% increase in the largest diameter of the lesion and stable disease - neither 30% decrease nor 20% increase of the largest diameter of the lesion.
  Change in the largest diameter:
Time Frame: 180 days after treatment
Population: There were 7 patients with a total of 44 cutaneous metastases which were randomized. We chose up to 10 tumours on each patient. At the first 6 tumours we examined the clinical response rate, and (if they had more) the rest 4 were used for biopsy. 33 from the 44 lesions were evaluated in clinical response, the rest were used for biopsy.
Measure: Number; unit: cutaneous metastases
Units Other Than Participants: cutaneous metastases
Groups:
- Calcium Electroporation: Volume of calcium chloride (220 mmol/L) was dependent on the tumor volume. Smaller tumors should have bigger volume per cm3, as smaller tumors were expected to have a bigger loss of injected medicine into the surrounding tissue. The dose volume was calculated according to the 'European Standard Operating Procedure of the Electrochemotherapi (ESOPE)'.
  * Tumor < 0.5 cm³ - 1 ml/cm³ tumor volume
  * Tumor > 0.5 cm³ - 0,5 ml/cm³ tumor volume Tumor volume = ab²π/6 (a = longest diameter, b = longest diameter perpendicular to "a")
  All patient's regardless of the number of metastases have had one biopsy from area treated with calcium and one from area treated with bleomycin, after the randomization code is revealed at day 180.
  All biopsies were handled according to current guidelines and analyzed by a pathologist for amount of tumor tissue, inflammation, fibrosis and necrosis.
- Bleomycin Based Electrochemotherapy: Both dose and volume of bleomycin (1000 IU/ml) is standard according to ESOPE.
  * Tumor < 0.5 cm³ - 1 ml/cm³ tumor volume
  * Tumor > 0.5 cm³ - 0,5 ml/cm³ tumor volume Tumor volume = ab²π/6 (a = longest diameter, b = longest diameter perpendicular to "a")
  Maximum of injected bleomycin per tumor was1500 IU and total dose per treatment 7500 IU. Normal maximum limit for bleomycin was 15.000 IU/m² body surface area.
  All patient's regardless of the number of metastases have had one biopsy from area treated with calcium and one from area treated with bleomycin, after the randomization code is revealed at day 180.
  All biopsies were handled according to current guidelines and analyzed by a pathologist for amount of tumor tissue, inflammation, fibrosis and necrosis.
Arm/Group | Calcium Electroporation | Bleomycin Based Electrochemotherapy
Number analyzed (Participants) | 7 | 7
Number analyzed (cutaneous metastases) | 18 | 15
cutaneous metastases
  CR | 4 | 6
  PR | 2 | 2
  SD | 6 | 5
  PD | 6 | 2
Statistical Analysis 1: Comparison: Calcium Electroporation vs Bleomycin Based Electrochemotherapy; After reviewing existing data from electrochemotherapy with intratumoral bleomycin on small cutaneous metastases ≤3cm , we estimated the expected response rate for electrochemotherapy to 85%. We have no clinical results for the treatment of calcium electroporation, but on the basis of preclinical studies, we decided to accept a difference in response of 20%. All statistical analysis were done using IBM SPSS v24; Test type: Non-Inferiority — Examined the objective response rate (ORR) that there was 20% difference between the 2 treatment arms at day 180. With a significance level of 0,05 and a power of 80% the study required 28 evaluable metastases; p = 0.30, Fisher Exact; Odds Ratio (OR) = 0.4489629, 95% CI 2-sided [-13.30 to 53.30]

2. Secondary Outcome: Adverse Events for Calcium Electroporation and Bleomycin Based Electrochemotherapy. The Adverse Reactions Are Classified According to CTCAE Version 4.0 (Common Terminology Criteria for Adverse Events).
Description: * Adverse Event, AE: Any adverse events in a patient that occur or worsen during the trial and does not necessarily have a causal relationship to study treatment
  * Adverse Reaction, AR: All noxious and unintended reactions to a trial drug at any dose (possible relation between the study drug and the adverse reaction cannot be excluded)
  * Unexpected Adverse Reaction, UAR: An adverse reaction with a nature or severity that is not in accordance with the current product information (Investigator's Brochure)
  * Serious Adverse Event, SAE: an event or side effect that at any dose:
  * Results in death
  * Is life threatening
  * Leads to hospitalization or prolongation of hospital stay
  * Results in persistent or significant disability or incapacity
  * Leads to a congenital anomaly or birth defect
  * Is a major medical event
  * Suspected Unexpected Serious Adverse Reactions, SUSARs: adverse reactions that are not described in the product information for the experimental drug
Time Frame: 180 days after treatment
Measure: Number; unit: cutaneous metastases
Units Other Than Participants: cutaneous metastases
Groups:
- Calcium Electroporation: Experiences from treating small tumors with electrochemotherapy, show that the treated area initially can become erythmatose and swollen, but this fades quickly. The area can then become necrotic which heals within 6-10 weeks. In a few cases, infection may occur in the treatment area. With calcium electroporation we expect to see the same response to treatment.
- Bleomycin Based Electrochemotherapy: At electrochemotherapy the most reported adverse events are pain after the procedure and flu-like symptoms. The latter is a reaction to bleomycin and is therefore not expected by calcium electroporation.
Arm/Group | Calcium Electroporation | Bleomycin Based Electrochemotherapy
Number analyzed (Participants) | 7 | 7
Number analyzed (cutaneous metastases) | 18 | 15
cutaneous metastases
  Ulceration | 2 | 3
  Hyperpigmentation | 2 | 6
  Flu-like symptoms | 0 | 0
  Itch | 0 | 0

3. Other Pre Specified Outcome: The Tertiary Outcome is to Register if Calcium Affects the Current Strength in Electroporation Treatments.
Description: We measured the maximum electric current which was given to the metastases. The measurement was needed because the current is unknown during Ca-electroporation, and also we would like to determine wether there is a difference between bleomycin based electrochemotherapy and calcium electroporation in current.
Time Frame: Day 0 - During Ca-electroporation and bleomycin based electrochemotherapy interventions
Measure: Median (Full Range); unit: Amper
Units Other Than Participants: cutaneous metastases
Groups:
- Calcium Electroporation: Calcium electroporation is a local treatment where calcium is administered intratumoral and followed by electrical pulses applied on the tumor. Volume of calcium chloride (220 mmol/L) was dependent on tumor volume which was calculated according to the 'European Standard Operating Procedure of the Electrochemotherapy' (ESOPE).
  Calcium chloride 220 mmol/L (9 mg/ml):
  * Tumor < 0,5 cm3 - 1 ml / cm3 tumor volume
  * Tumor >0,5 cm3 - 0,5 ml/ cm3 tumor volume Tumor volume = ab2π/6 (a=longest diameter, b= longest diameter perpendicular to a)
- Bleomycin Based Electrochemotherapy: Electroporation is a method that can facilitate transport of molecules across the cell membrane and into the cell by means of electrical pulses. The method can be used with molecules that normally have difficulty passing the cell membrane such as chemotherapy (electrochemotherapy).The most used chemotherapeutic drug used in electrochemotherapy is bleomycin (1000 IU/ml). Both dose and volume of bleomycin is standard according to ESOPE.
  Bleomycin 1000 IU/ml:
  * Tumor < 0.5 cm³ - 1 ml/cm³ tumor volume
  * Tumor > 0.5 cm³ - 0,5 ml/cm³ tumor volume Tumor volume = ab²π/6 (a = longest diameter, b = longest diameter perpendicular to "a")
  Maximum of injected bleomycin per tumor was 1500 IU and total dose per treatment was 7500 IU.
Arm/Group | Calcium Electroporation | Bleomycin Based Electrochemotherapy
Number analyzed (Participants) | 7 | 7
Number analyzed (cutaneous metastases) | 18 | 15
Amper | 3.850 [1.400 to 9.000] | 4.000 [1.400 to 6.500]

ADVERSE EVENTS:
Time Frame: 180 days after treatment
Description: Any adverse events in a patient that occur or worsen during the trial and does not necessarily have a causal relationship to study treatment
Arm/Group | Calcium Electroporation | Bleomycin Based Electrochemotherapy
All-Cause Mortality (participants affected / at risk) | 1/7 | 1/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 1/7 | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Calcium Electroporation (N=7) | Bleomycin Based Electrochemotherapy (N=7)
Other primary tumor (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
The study has certain limitations, like the small number of enrolled metastases, and the use of different electrodes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/17/NCT03628417/Prot_SAP_000.pdf